CLINICAL TRIAL: NCT06843135
Title: Synchrony in Cardiac Conduction: Assessing the Effects of Pacing on Cardiac Performance Through Magnetic Resonance Imaging and Advanced ECG-imaging
Acronym: HARMONY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Luuk Hopman, Postdoctoral Research Fellow, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL88751.018.25
Record Dates: First submitted 2025-02-02; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; AV Block
MeSH Terms: conditions — Heart Failure; Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conduction system pacing (Active Comparator)
  Interventions: Device: Ventricular pacing
- Right ventricular pacing (Active Comparator)
  Interventions: Device: Ventricular pacing

INTERVENTIONS:
Device: Ventricular pacing — Participants will undergo conductionsystem pacing and right ventricular pacing in a randomized sequence, each for six months. After each phase, patients will undergo a CMR scan and advanced ECG imaging

SUMMARY:
Rationale Right ventricular pacing (RVP) is an established and effective therapy for patients with atrioventricular (AV) block. However, frequent RVP has been associated with left ventricular (LV) dyssynchrony and may progess heart failure. Conduction system pacing (CSP), a recently introduced alternative to RVP, aims to preserve physiological ventricular activation by engaging the heart's native conduction system. CSP includes diverse pacing approaches such as selective or non-selective His-bundle pacing, selective left bundle pacing, and LV-septal pacing, each with varying levels of fidelity in reproducing normal conduction. The mechanical impact of these distinct CSP strategies on left and right ventricular (RV) performance remains poorly understood.

Cardiac magnetic resonance imaging (CMR), a non-invasive and highly accurate tool for assessing cardiac structure and function, is uniquely positioned to elucidate the effects of CSP and RVP on cardiac performance. This trial aims to evaluate the comparative mechanical effects of these pacing strategies, potentially identifying the optimal approach for improving outcomes in patients with AV block.

Objective To investigate and compare the effects of CSP and RVP on cardiac performance, as assessed by CMR and electrocardiographic imaging (ECG-imaging).

Main Trial Endpoints The primary endpoints are measures of LV and RV performance assessed via CMR, including: ventricular volumes, ejection fraction (EF), and myocardial strain

Secondary Trial Endpoints

Secondary endpoints include:

Safety and Feasibility:

* Adverse events (e.g., troponin release, lead displacement, arrhythmias, heart failure).
* Technical feasibility (e.g., ease of device implantation, ability to maintain proper pacing).

Electrophysiological Assessment:

* Degree of selectivity in engaging the native conduction system.
* Ventricular activation times as assessed by ECG-imaging.

Trial Design This is a randomized, controlled, single blind, two-center crossover trial. Participants will undergo CSP and RVP in a randomized sequence, each for six months. CMR and ECG-imaging will be performed at 6 months (end of the first pacing phase) and 12 months (end of the second pacing phase).

Trial Population The trial will enroll 88 patients with a normal of at most mildly reduced ejection fraction and an indication for ventricular pacing.

Interventions Participants will undergo CMR and ECG-imaging at 6 months and 12 months.

Ethical Considerations This trial is designed to advance understanding of the mechanical and clinical effects of CSP relative to RVP in patients with AV block. The anticipated benefits include improved cardiac performance and enhanced quality of life. The primary burden to participants is the requirement for an additional CMR scan, which may be perceived as inconvenient or even stressful. The trial minimizes risk by utilizing established clinical procedures and closely monitoring participants for adverse events.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age ≥ 18 years
* Patients with a left ventricular ejection fraction of ≥35%
* Patients with an indication for ventricular pacing and high-degree atrioventricular block where the degree of anticipated RV pacing is >20% including:
* Third degree AV block
* Symptomatic or asymptomatic second-degree AV block
* High degree AV block
* Pace and ablate (AV-node ablation)

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* CRT indication (patients with heart failure (NYHA >1) in sinus rhythm with left ventricular ejection fraction (LVEF) <35%, QRS duration >150 ms, and left bundle branch block (LBBB) QRS morphology despite optimised medical therapy)
* Inability to undergo CMR (i.e. severe claustrophobia or MRI contraindications)
* Life expectancy <12 months
* Indication for an implantable cardioverter defibrillator
* Presence of severe valve disease or mechanical valves
* Any prior attempt at implantation of an ICD, CRT, CSP
* Permanent AF with rapid ventricular response, unless pace and ablate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is LV ejection fraction measured on CMR | At 6 months after crossover

IPD SHARING:
Plan to Share IPD: Undecided